CLINICAL TRIAL: NCT04843891
Title: Preliminary Evaluation of [64Cu] Macrin in Healthy Individuals and Subjects With Cardiovascular Disease, Sarcoidosis and Malignancy.
Brief Title: Evaluation of PET Probe [64]Cu-Macrin in Cardiovascular Disease, Cancer and Sarcoidosis.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ralph Weissleder, MD (Other)
Responsible Party: Sponsor-Investigator, Ralph Weissleder, MD, Professor of Radiology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021P000355
Record Dates: First submitted 2021-03-31; First posted 2021-04-14 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Sarcoid; Cardiovascular Diseases; Cancer
MeSH Terms: conditions — Sarcoidosis; Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible subjects, including healthy volunteers and patients with sarcoidosis, cardiovascular disease and cancer, will be enrolled to undergo imaging with the PET Probe [64]Cu Macrin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healthy Volunteers (Experimental): In 10 healthy volunteers the radiation dosimetry, normal organ distribution, and safety of [64Cu]-Macrin injection will be studied.
  Interventions: Drug: [64]Cu Macrin
- Cardiovascular Disease (Experimental): In 30 subjects with a history of recent myocardial infarct, the radiation dosimetry, normal organ distribution, and safety of [64Cu]-Macrin injection will be studied. In addition, the ability of [64Cu] Macrin to concentrate at the infarct site will be correlated with cardiac MRI.
  Interventions: Drug: [64]Cu Macrin
- Cancer (Experimental): In 30 subjects with an epithelial malignancy the radiation dosimetry, normal organ distribution, and safety of [64Cu]-Macrin injection will be studied. In addition, the ability of [64Cu] Macrin to concentrate at the tumor site will be correlated with imaging and histopathology, where available.
  Interventions: Drug: [64]Cu Macrin
- Sarcoidosis (Experimental): In 30 subjects with sarcoidosis the radiation dosimetry, normal organ distribution, and safety of [64Cu]-Macrin injection will be studied. In addition, the ability of [64Cu] Macrin to concentrate at the tumor site will be correlated with imaging and histopathology, where available.
  Interventions: Drug: [64]Cu Macrin

INTERVENTIONS:
Drug: [64]Cu Macrin — Up to 15 mCi of [68Ga]CBP8 will be administered to each subject.

SUMMARY:
To evaluate the safety of [64Cu] Macrin and its whole-body distribution, metabolism, pharmacokinetics, and radiation burden in healthy volunteers. To detect [64Cu]-Macrin accumulation in sites of disease in subjects with cancer, sarcoidosis or myocardial infarct.

DETAILED DESCRIPTION:
Macrophages are phagocytic cells of the innate immune system. Their accumulation is a hallmark of many inflammatory diseases and they have diverse roles in tissue responses to infection and injury and in tissue repair. As macrophages have a tissue specific and often disease stage specific roles, future therapies directed at macrophage subtypes at certain points in the course of a disease may be more efficacious and result in less systemic side effects, as compared to conventional chemotherapeutics. [64Cu] Macrin is designed to detect macrophages by PET imaging. As a result, PET imaging can be used to identify inflammatory "hotspots" and quantitate local macrophage density non-invasively. The investigators studies in mice showed that [64Cu] Macrin has excellent pharmacological and pharmacokinetic profile with high target uptake and low retention in background tissues and organs.

The investigators wish to first evaluate in healthy human subjects the pharmacological and pharmacokinetic profile, and the overall safety of the new radiopharmaceutical [64Cu] Macrin. The investigators will then establish the concentration of [64Cu] Macrin in patients following myocardial infarct, in sarcoidosis and in cancer patients. In a subset of patients where tissue sampling is feasible, we will correlate tracer uptake on imaging to macrophage density on histopathology or with additional standard of care imaging studies.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Healthy subjects

* Must be 18 years of age or older
* Must be deemed healthy at screening visit, as determined by the physician investigator or nurse practitioner, based on the following assessments at screening: physical examination, medical history and vital signs;

  * No known history of pre-existing cardiac or respiratory disease or malignancy
  * Have the ability to give written informed consent.

Group 2: Myocardial Infarction

* History of percutaneous coronary intervention (PCI) for acute or chronic coronary syndrome (within 3-5 days)
* Have the ability to give written informed consent
* Must be 18 years of age or older
* Hemodynamically stable

Group 3: Sarcoidosis

* A suspected or confirmed diagnosis of intrathoracic sarcoidosis
* Have the ability to give written informed consent
* Must be 18 years of age or older

Group 4: Malignancy

* Suspected or confirmed thoracic, intra-abdominal or pelvic malignancy
* Have the ability to give written informed consent
* Must be 18 years of age or older

Exclusion Criteria:

* • Electrical implants, such as cardiac pacemaker or perfusion pump;

  * Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, metallic tattoos anywhere on the body, tattoos near the eye, or steel implants ferromagnetic objects such as jewelry or metal clips in clothing;
  * eGFR of less than 30 mL/min/1.73 m2 within the past 30 days;
  * Pregnant or breastfeeding (a negative quantitative serum hCG pregnancy test is required for females having child-bearing potential before the subject can participate);
  * Self-reported or documented claustrophobic reactions;
  * Research-related radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months);
  * Unable to lie comfortably on a bed inside the MR-PET;
  * BMI > 33 (limit of the PET-MRI table);
  * Determined by the investigator(s) to be clinically unsuitable for the study (e.g. based on screening visit and/or during study procedures);
  * Stroke within the last 3 months;
  * Cardiac or major surgery within the last 3 months;
  * History of abnormal heart rate including persistent tachyarrhythmia (heart rate persistently >120 bpm) or bradyarrhythmia (heart rate persistently < 50 bpm);
  * History of atrial premature complexes with daytime pauses > 3s;
  * Contraindications to gadolinium-based contrast agents, including an eGFR < 30 mL/min (myocardial infarction and sarcoidosis patients only).
  * History of myeloproliferative disorder.
  * Age >80 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-04-05 (Estimated)

PRIMARY OUTCOMES:
To establish human dosimetry of 64Cu Macrin in Healthy Volunteers | 1 year
  We will use established methods to provide quantitative information on the amount of [64Cu] Macrin radioactivity that accumulates in peripheral organs and brain. Dose-corrected imaging data will be processed using time-activity curves based on ROIs manually-drawn on MR data and projected onto PET datasets.
[64Cu] Macrin accumulation and detection in cancer | 1 year
  Probe uptake will be measured in organs affected by solid epithelial malignancies and compared to uptake in the uninvolved parts of the organs and in these organs in healthy volunteers. We expect greater uptake in the part of the organs affected by malignancy.
[64Cu] Macrin accumulation and detection in myocardial infarction | 1 year
  Probe uptake will be measured at a myocardial infarct and compared to uptake in the remainder of the heart and in the hearts of healthy volunteers. We expect greater uptake at the site of a myocardial infarction.
[64Cu] Macrin accumulation and detection in sarcoidosis | 1 year
  Probe uptake will be measured in the heart and lungs of patients with sarcoidosis and compared to uptake in these organs in healthy volunteers. We expect greater uptake in the organs affected by sarcoidosis.

SECONDARY OUTCOMES:
[64Cu] Macrin accuracy for macrophage localization | 1 year
  To determine the sensitivity and specificity of [64 Cu] Macrin accumulation for the detection at sites of inflammation by comparing tracer accumulation to histopathology and/or standard of care imaging studies

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Aileen O'Shea, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No